CLINICAL TRIAL: NCT06310317
Title: Evaluating the Effect of Use of Technologies to Increase the Cognitive Abilities in Children With Autism Spectrum Disorders
Brief Title: Applied Behavior Analysis With Technologies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Responsible Party: Principal Investigator, Flavia Marino, Head of Unit, Istituto per la Ricerca e l'Innovazione Biomedica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNR-IRIB-PRO-2024-003
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Autism; Autism Spectrum Disorder
Keywords: Autism; autism spectrum disorder; children; Applied Behavior Analysis; ABA
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): 15 children belonging to the experimental group will undergo the treatment carries out the procedure by means of stimuli presented with technologies supports
  Interventions: Behavioral: Applied Behavior Analysis protocol
- control group (Other): 15 children belonging to the control group will undergo the treatment by performing the procedure with images printed on laminated A4 sheets.
  Interventions: Behavioral: Traditional intervention

INTERVENTIONS:
Behavioral: Applied Behavior Analysis protocol — The main objective of the experimental protocol is to promote the development of cognitive skills, facilitate the acquisition of new skills and promote the adoption of functional and adaptive behaviors. The use of Applied Behavior Analysis procedures, with the help of technological tools such as a tablet or robot can facilitate the increase of new knowledge and skills.
  The criterion is acquired if the subject emits 8 out of 10 independent correct responses (90%) for 3 consecutive sessions.
  The objective is to test whether the technological tool used (tablet or robot) can make the proposed learning procedure more effective. The experimental group carries out the procedure by means of stimuli presented on tablets or robots.
  Arms: experimental group
Behavioral: Traditional intervention — The main objective of the experimental protocol is to promote the development of cognitive skills, facilitate the acquisition of new skills and promote the adoption of functional and adaptive behaviors. In this group the materials are traditional, such as image printed. The criterion is acquired if the subject emits 9 out of 10 independent correct responses (90%) for 3 consecutive sessions. The control group performs the procedure with images printed on A4 laminated sheets.
  Arms: control group

SUMMARY:
Applied Behavior Analysis (ABA) is a therapeutic approach for autism that is based on the principles of behavioral theory, learning, and positive reinforcement. Current research shows that early and intensive ABA intervention is effective in reducing dysfunctional behaviors and promoting learning and enactment of socially appropriate behaviors.

In this context, new approaches that attempt to integrate advanced technologies can play a key role. This experimental protocol aims to test whether the use of advanced technologies, such as tablets, as part of an intervention for a group of children with autism spectrum disorder (ASD) is more effective than the traditional approach implemented in a control group of children with ASD. The experimental protocol is aimed at enhancing cognitive skills, increasing new skills and acquiring functional/adaptive behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Children with diagnosis of autism

Exclusion Criteria:

* presence of other medical disorders

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Verbal Behavior Milestones Assessment and Placement Program (VB-MAPP) | the test need approximately 1 hour
  Is an assessment tool that attends to all those skills that are fundamental to the development and enhancement of verbal communication skills and the proper use of language in social interactions. It focuses especially on the assessment of language prerequisites fundamental to the development of verbal behavior in accordance with the classification of verbal operants proposed by Skinner: mand, tact, echoic, intraverbal. It consists of a manual, a protocol and a set of materials (pictures and standardized items for assessment). The protocol is divided into:
  * Tables
  * Early Echoic Skills Assessment (EESA) - Assessment of barriers: behaviors that might hinder the child's learning
  * Assessment of transitions: the child's ability to make the transition to teaching modes based on the natural context
  * Task Analysis and Skills Monitoring: describes the individual milestones required to reach the main milestone
  * Scoring grids

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Marino, Principal Investigator — Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR)
Locations (1):
- Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR), Messina, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi KR, Bhakta B, Knight EA, Becerra-Culqui TA, Gahre TL, Zima B, Coleman KJ. Patient Outcomes After Applied Behavior Analysis for Autism Spectrum Disorder. J Dev Behav Pediatr. 2022 Jan 1;43(1):9-16. doi: 10.1097/DBP.0000000000000995. PMID 34342287
- [Background] Yu Q, Li E, Li L, Liang W. Efficacy of Interventions Based on Applied Behavior Analysis for Autism Spectrum Disorder: A Meta-Analysis. Psychiatry Investig. 2020 May;17(5):432-443. doi: 10.30773/pi.2019.0229. Epub 2020 May 8. PMID 32375461
- [Background] Valencia K, Rusu C, Quinones D, Jamet E. The Impact of Technology on People with Autism Spectrum Disorder: A Systematic Literature Review. Sensors (Basel). 2019 Oct 16;19(20):4485. doi: 10.3390/s19204485. PMID 31623200